CLINICAL TRIAL: NCT03967431
Title: Effects of Narrative Enhancement and Cognitive Therapy (NECT) on Self-stigma in Patients With Schizophrenia: A Randomized Controlled Study
Brief Title: Effects of Narrative Enhancement and Cognitive Therapy (NECT) on Self-stigma in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB1070910-02
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2019-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The participants were divided into experimental and control groups through block randomization.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrative Enhancement and Cognitive Therapy group (Experimental): The patients in the experimental group received narrative enhancement and cognitive therapy which contains 20 times group meetings.
  Interventions: Other: Narrative Enhancement and Cognitive Therapy (NECT)
- Control group (No Intervention): The patients in the control group received routine care.

INTERVENTIONS:
Other: Narrative Enhancement and Cognitive Therapy (NECT) — Narrative Enhancement and Cognitive Therapy includes two introduction meetings, three psychoeducation meetings, seven cognitive restructuring meetings, seven narrative enhancement meetings and one summing up meeting.
  Arms: Narrative Enhancement and Cognitive Therapy group

SUMMARY:
This study aims to explore the effect of narrative enhancement and cognitive therapy in improving self-stigma, self-esteem, depression and hope of patients with chronic schizophrenia.

DETAILED DESCRIPTION:
86 participants with chronic schizophrenia in two different hospitals in northern Taiwan were recruited in this study. All participants were randomized into experimental and control groups through block randomization. After randomization, the participants in control group received routine care and the others in experimental group received Narrative Enhancement and Cognitive Therapy(NECT) which contains 20 times group meetings. The research tools include demographic data, the Internalized Stigma of Mental Illness Scale (ISMIS), the Discrimination and Stigma Scale (DISC), Rosenberg self-Esteem scale (RSES), Beck Depression Inventory (BDI-II) and Herth Hope Index (HHI). The questionnaires were collected for three times, including before the intervention, 12 weeks after intervention, and after the end of intervention. The collected data were analyzed by IBM SPSS 24.0 statistical software. The descriptive statistics include mean, standard deviation, minimum, maximum, frequency distribution, and percentages; the Generalized estimating equations (GEE) were used to explore the effect of Narrative Enhancement and Cognitive Therapy on self-stigma, self-esteem, depressive symptoms and hope in patients with schizophrenia after controlling demographic data.

ELIGIBILITY:
Inclusion Criteria:

* People with Schizophrenia for more than two years.
* The age is between 20(included) and 64(included).
* Can communicate with Mandarin or Taiwanese.
* The score of the Mini-Mental State Examination (MMSE) is above 24(included).
* The score of the Positive and Negative Syndrome Scale(PANSS) is below 60(included).
* People are willing to participate in this study, can read and know the consent and can sign on the consent by their own.

Exclusion Criteria:

* Exclude people with a personality disorder, brain injury, cognitive impairment, Intellectual Developmental Disorder or substance use disorder.
* people who are not willing to sign the consent.
* people can not read.
* people can not communicate with Mandarin or Taiwanese.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
The Internalized Stigma of Mental Illness Scale (ISMIS) | For two groups at baseline(T0), at 12th week(T1) and at 20th week(T2)
  To measure internalized stigma. There are five sub-scales in ISMIS, including Alienation(6 items), Stereotype Experience(7 items), Discrimination Experience(5 items), Social Withdrawal(6 items) and Stigma Resistance(5 items). There are 29 items in this scale. Using Likert scale to rate each item (1=Strongly disagree, 2=disagree, 3=agree, 4=strongly agree) and higher score means higher internalized stigma.
The Discrimination and Stigma Scale | For two groups at baseline(T0), at 12th week(T1) and at 20th week(T2)
  To know the experiences of discrimination and stigma. There are four sub-scales in DISC, including Unfair Treatment, Stopping Self, Overcoming Stigma and Positive Treatment. These four sub-scales are independent. Using four point to rate each item(0=not at all, 1=a little, 2=Moderately, 3=A lot) or choose "Not applicable" if the item is not applicable for the subject.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI-II) | For two groups at baseline(T0), at 12th week(T1) and at 20th week(T2)
  To know the level of depressive symptoms.There are 21 items in BDI-II. Using 0 to 3 to rate each item. The higher score a participant get, a higher depressive symptoms a participant has.
Herth Hope Index (HHI) | For two groups at baseline(T0), at 12th week(T1) and at 20th week(T2)
  To measure the level of hope. There are 12 items in this scale. Using Likert scale to rate each item (1=Strongly disagree, 2=disagree, 3=agree, 4=strongly agree) and higher score means higher level of hope.
Rosenberg self-esteem scale | For two groups at baseline(T0), at 12th week(T1) and at 20th week(T2)
  To measure the level of self-esteem.There are 10 items in this scale. Using Likert scale to rate each item (1=Strongly disagree, 2=disagree, 3=agree, 4=strongly agree) and higher score means higher level of self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Chiu-Yueh Yang, Ph.D., Study Chair — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No